CLINICAL TRIAL: NCT01461434
Title: Randomized Controlled Trial to Evaluate Implanted Event Recorders for the First Diagnosis of Atrial Fibrillation in High-risk Patients
Brief Title: Graz Study on the Risk of Atrial Fibrillation
Acronym: GRAF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Frank R Heinzel, MD, PhD, Associate Professor Frank R. Heinzel, MD, PhD, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GRAF-01-SCCT
Record Dates: First submitted 2011-10-23; First posted 2011-10-28 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Atrial Fibrillation; Hypertension; Diabetes; Chronic Heart Failure; Vascular Disease
Keywords: atrial fibrillation; biomarkers; stroke prevention; implantable loop recorder
MeSH Terms: conditions — Atrial Fibrillation; Hypertension; Diabetes Mellitus; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- loop recorder (Experimental): patients will be implanted with a subcutaneous loop recorder and have regular follow-ups
  Interventions: Device: Medtronic Reveal XT implantable loop recorder
- regular follow-up (No Intervention): patients will receive regular follow-ups with standard ECG

INTERVENTIONS:
Device: Medtronic Reveal XT implantable loop recorder — subcutaneous implantation
  Arms: loop recorder

SUMMARY:
Atrial fibrillation (AF) is the most common clinical arrhythmia. AF is associated with increased risk for stroke due to blood clots formed in the fibrillating atria. Some patient characteristics increase the likelyhood of AF and at the same time the risk of stroke when AF has developed. To reduce the risk of stroke, anticoagulation therapy is recommended in patients with AF and risk factors (such as high blood pressure, diabetes, vessel disease). However, occasional (paroxysmal) AF may occur without symptoms and remain undetected, leaving patients at risk.

Aim of the prospective randomized study is to compare two management strategies for patients at increased risk for AF but without a known history of AF. Patients are seen regularly (monthly, then quarterly) for follow-up (incl. ECG recording and blood sample). One group of patients additionally receives a subcutaneous implantation of a loop recorder for continuous rhythm monitoring, while the control group remains on standard follow-up. Observation period is one year (optional extension for 3 years). The time to first diagnosis of AF is compared between groups, blood samples are analyzed for potential biomarkers of AF.

ELIGIBILITY:
Inclusion Criteria:

* CHA2DS2-VASc risk score >= 4*
* 18 years or older

Exclusion Criteria:

* known history of atrial fibrillation
* implanted rhythm device
* pre-existing indication for oral anticoagulation

(*)CHA2DS2-VASc: C - chronic heart failure (1 point); H - hypertension (1 point); A - age >= 75 years (2 points); D - diabetes (1 point); S - stroke (2 points); V - vascular disease (1 point); A - age >=65 and < 75 years (1 point); Sc - sex category (female) (1 point) ;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-11; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Time to first diagnosis of atrial fibrillation | 12 months

SECONDARY OUTCOMES:
Time to change in therapy based on the diagnosis of atrial fibrillation | Baseline (0 months), 1,2,3,4,5,6,9 and 12 months
Hospitalizations | 12 months
Change in NTproBNP serum level associated with occurrence of atrial fibrillation | Baseline (0 months), 1,2,3,4,5,6,9 and 12 months
Death | 12 months
Stroke | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- LKH/Uniklinikum - Klinische Abteilung für Kardiologie, Graz, Austria